CLINICAL TRIAL: NCT06287073
Title: A Regulatory Non-interventional Study to Monitor the Safety and Efficacy of JARDIANCE® (Empagliflozin 10 mg) in Korean Patients With Chronic Kidney Disease (CKD)
Brief Title: JARDIANCE® Post Marketing Surveillance in Korean Patients With Chronic Kidney Disease (CKD)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0323; EUPAS107293 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2024-02-23; First posted 2024-02-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- New JARDIANCE® users with chronic kidney disease (CKD): Patients with CKD starting JARDIANCE® for the first time in accordance with the approved label in Korea
  Interventions: Drug: JARDIANCE®

INTERVENTIONS:
Drug: JARDIANCE® — JARDIANCE®

SUMMARY:
The primary objective is to monitor the safety profile of JARDIANCE® in Korean patient with chronic kidney disease (CKD) in routine clinical practice.

The secondary objective is to monitor the efficacy of JARDIANCE® by evaluating changes in urine albumin-creatinine ratio (UACR) after 12 and/or 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧19 years at enrolment
* Patients diagnosed with CKD
* Patients with CKD starting JARDIANCE® for the first time in accordance with the approved label in Korea
* Patients who have provided informed consent and signed the data release consent form

Exclusion Criteria:

* Patients with previous exposure to JARDIANCE®
* Patients with hypersensitivity to empagliflozin or to any of the excipients
* Patients with type 1 diabetes
* Patients with history of Diabetic Ketoacidosis (DKA)
* Patients with rare hereditary conditions of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
* Patients who are pregnant or are breastfeeding or who plan to become pregnant during the study period

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single-arm, open-label, multi-centre observational and non-interventional study (ONIS) based on newly collected data. This study will be carried out by enrolling patients in a consecutive manner into the study requiring completion of case report forms (CRFs) for all participants who initially administered JARDIANCE® following the study start date until the planned number of participants is reached.
Sampling Method: Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Up to 24 weeks
Number of subjects with serious adverse event | Up to 24 weeks
Number of subjects with non-serious adverse events | Up to 24 weeks
Number of subjects with adverse drug reaction | Up to 24 weeks
Number of subjects with serious adverse drug reactions | Up to 24 weeks
Number of subjects with unexpected adverse events | Up to 24 weeks
Number of subjects with adverse events of special interest | Up to 24 weeks
  Adverse events of special interest are: liver injury, ketoacidosis in diabetic and nondiabetic population, lower limb amputation
Number of subjects with specific adverse events | Up to 24 weeks
  Specific adverse events are: severe hypoglycaemia, urinary tract infection, genital infection, bone fracture, urinary tract malignancy, volume depletion, acute kidney injury, gout, hyperkalaemia
Number of subjects with adverse events leading to temporary or permanent discontinuation | Up to 24 weeks
Number of subjects with adverse events by intensity | Up to 24 weeks
  Intensity is measured as: mild, moderate, severe
Number of subjects with adverse events by outcome of the events | Up to 24 weeks
  Outcome of the event is measured as: recovered, not yet recovered, sequela, fatal, unknown
Number of subjects with adverse events by causality | Up to 24 weeks
  Causality is measured as: certain, probable·likely, possible, unlikely, conditional· unclassified, unassessable·unclassifiable
Number of subjects with adverse events leading to death | Up to 24 weeks

SECONDARY OUTCOMES:
Occurrence of change in urine albumin-creatinine ratio (UACR) from baseline after 12 weeks and/or 24 weeks of treatment | at baseline, at Week 12, and at Week 24

CONTACTS AND LOCATIONS:
Locations (12):
- South Korea (12):
  - Hallym University Sacred Heart Hospital, Anyang
  - Chungbuk National University Hospital, Cheongiu
  - Yonsei University Wonju Severance Christian Hospital, Gangwon
  - Inje University Ilsan Paik Hospital, Goyang
  - Chonnam National University Hospital, Gwangju
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Soonchunhyang University Hospital Seoul, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Yeouido St.Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame frame' are fulfilled , researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents upon signing of a 'Document Sharing Agreement'. For study data 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com